CLINICAL TRIAL: NCT03343691
Title: Blood Test for Early Detection of Breast Cancer Using Todos Medical -Breast 1(TM-B1) Assay
Acronym: TM-B1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Todos Medical, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IL-TM-B1-01
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect blood from the subject in two 6 ml K2 EDTA blood collection tube (total 12 ml blood) according to standardized phlebotomy procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening Population: Cohort 1:Screening Population - Women presenting for routine XRM and / or breast US.
  Participants will be followed for one year and the outcome of those who undergo an annual XRM / breast ultrasound will be recorded.
  Interventions: Diagnostic Test: Screening Population
- Breast Cancer Population: Cohort 2:Breast Cancer Population - Women who were diagnosed with malignant breast tumors, as determined by biopsy, and have not yet begun any treatment for the disease.
  Interventions: Diagnostic Test: Breast Cancer Population

INTERVENTIONS:
Diagnostic Test: Screening Population — Blood samples taken from screening population
  Groups: Screening Population
Diagnostic Test: Breast Cancer Population — Blood samples taken from Breast Cancer population
  Groups: Breast Cancer Population

SUMMARY:
Blood samples from a total of 200 women in two cohorts will be collected and analyzed by TM-B1 assay, which is based on TBIA (Total Biochemical Infrared Analysis) to confirm the presence of cancer. These two cohorts will yield 75 healthy women with no pathological findings, 75 women diagnosed as having benign breast tumor and 50 women diagnosed as having breast cancer.

DETAILED DESCRIPTION:
Prospective, two arms, observational, blinded, cohort study enrolling 200 women which intended to validate the cut-off points between women with malignant tumors, benign tumors, and women without tumors (controls) and to validate the sensitivity and specificity of TM-B1 for the detection of an invasive breast tumor.

Two cohorts will be tested with TM-B1. The cohorts will differ in the percentage of women that are expected to yield a positive finding for breast cancer. Any finding in TM-B1 will not influence medical standards of care.

ELIGIBILITY:
Inclusion Criteria:

Screening Population:

* Subject signed the informed consent.
* Subject is aged 25 years and older.
* Subject is presenting for routine screening or diagnostic XRM and / or breast US.

Breast Cancer Population

* Subject signed the informed consent form.
* Subject is aged 25 years and older.
* Subject was diagnosed with a malignant breast tumor, and has not yet started treatment.

Exclusion Criteria:

All Subjects:

* Subject has been diagnosed with any type of malignancy apart from breast cancer.
* Subject has been previously treated for breast cancer.
* Subject underwent any surgery within the previous year (apart from benign nevus removal).
* Subject was treated for benign tumor within the previous year (e.g. polyps or cysts).
* Subject has an active infection or inflammation from any type of infection (bacterial or viral) as determined clinically at screening.
* Subject is currently taking medications related directly to, or that can affect, the immune system such as steroids.
* Subject has any type of active autoimmune disease such as lupus or rheumatoid arthritis.
* Diagnostic drugs (e.g. contrast materials) were injected or given orally to subject within the last 7 days prior to sample collection for TM-B1 analysis.
* Subject has been taking any investigational drug which influence her health status within 30 days prior to sample collection for TM-B1 analysis.
* Subject is not feeling well at the time of blood collection for TM-B1 analysis due to suspected bacterial or viral infection or subject has symptoms such as high fever, diarrhea, headache, vomiting, dizziness etc.
* Subject is pregnant, lactating, or undergoing fertility treatment.
* Subject has participated in this study, in another cohort, and the TM-B1 test was performed.

Breast Cancer Population only:

* The subject's tumor has been surgically removed before sample collection for TM-B1 analysis.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing a breast biopsy or a screening mammography,
Study Population: Cohort 1: Screening Population - Women presenting for routine XRM and / or breast US.
  Cohort 2: Breast Cancer Population - Women who were diagnosed with malignant breast tumors, as determined by biopsy, and have not yet begun any treatment for the disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
This study is intended to evaluate the sensitivity and specificity of the TM-B1 test compared to the Gold Standard diagnostic methods and clinical evaluations based on Digital X-Ray Mammography (XRM), and / or ultrasound, and / or MRI and / or pathology. | Timepoint 1, day 1
  the subject's blood (Groups 1 and 2)will be tested for the presence of breast cancer

SECONDARY OUTCOMES:
For asymptomatic women who have dense breast tissue (parenchymal density > 50% on XRM), evaluate the performance, in terms of sensitivity and specificity, of the TM-B1 test and XRM together as a breast cancer screening procedure compared to the XRM alone | Timepoint one, day 1
  The subject's blood (Groups 1 and 2) will be tested for the presence of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Tanir N Alweis, M.D., Principal Investigator — Kaplan Medical Center,Pasternak St., POB 1, Rehovot 76100, Israel
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No